CLINICAL TRIAL: NCT02058420
Title: Effect of Tocotrienols on Bone Health: A Pilot Study
Brief Title: Tocotrienols and Bone Health of Postmenopausal Women
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center (Other)
Collaborators: Texas Woman's University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB L14-056; American River Nutrition (Other: ARN)
Record Dates: First submitted 2014-02-01; First posted 2014-02-10 (Estimated); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Osteoporosis
Keywords: bone health
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo group (No Intervention): No active dose of tocotrienols
- Low tocotrienols group (Active Comparator): Low dose of tocotrienols
  Interventions: Drug: Low tocotrienols group
- High tocotrienols group (Active Comparator): High dose of tocotrienol
  Interventions: Drug: High tocotrienols group

INTERVENTIONS:
Drug: Low tocotrienols group — 300 mg tocotrienols daily
  Arms: Low tocotrienols group
Drug: High tocotrienols group — 600 mg tocotrienols daily
  Arms: High tocotrienols group

SUMMARY:
Osteoporosis (severe bone loss) is a bone disease with bone fragility and an increased chance for bone fractures. Women are 4 times more likely to have osteoporosis than men because there is no estrogen protection after menopause and women in general have lighter and thinner bones. Recent studies have indicated tocotrienols (one kind of vitamin E) supplement may be good for the bone health in postmenopausal women. However, no study has ever been done the role of tocotrienols in bone health in postmenopausal women. Our long-term goal is to develop a new strategy featuring a dietary supplement (i.e., tocotrienols) for slowing down bone loss in postmenopausal women. The purpose of the study is to examine the effect of 12-week tocotrienols on bone measurements in postmenopausal women. Investigators plan to recruit postmenopausal women using flyers, non-solicited e-mail system, campus announcement, local radio, newspapers, and TV scripts. We plan to enroll approximately 200 women to obtain 78 qualified women at the start of the study. After screening, qualified participants will be matched by body weight and age, and then randomly assigned to no tocotrienols, low tocotrienols, or high tocotrienols group. The outcome measures will be assessed at baseline, after 6, and after 12 weeks. Bone-related measurements will be recorded using blood and urine samples. Investigators will monitor safety of subjects after 6 and after 12 weeks. Food intake, physical activity, and quality of life will be assessed at baseline and 12 weeks. All data will be analyzed statistically.

ELIGIBILITY:
Inclusion criteria

1. Postmenopausal women with no menses for 1-10 years.
2. Bone mass with bone mineral density (BMD) T-score between 0.5 and -2.5 at the spine and/or hip.
3. Normal laboratory evaluation, thyroid function: TSH > 0.3 and < 5.0 mU/L; hepatic function: bilirubin ≤ 2.0 mg/dl; SGOT (also called AST)/SGPT (also called ALT) < 3x upper limit of normal; renal function: serum creatinine ≤ 2.0 mg/dl; BUN less than 1.5 times upper limit of normal; serum calcium, phosphorus, and alkaline phosphatase: within normal ranges. HbA1c < 7.0%.
4. Serum 25-OH vitamin D >= 20 ng/mL.
5. Age 40 and older

Exclusion criteria

1. History of, or evidence for, metabolic bone disease including recent fractures (other than low BMD).
2. Having received medication (calcitonin, raloxifene, or systemic glucocorticoids) within 3 months before the start of the study.
3. Having bisphosphonate within 12 months before the start of the study.
4. Having hormone/hormone-like replacement therapy within 3 months before the initiation of the study.
5. History of cancer except for treated superficial basal or squamous cell carcinoma of the skin.
6. History or evidence of endocrine disease or malabsorption syndrome that would be a contraindication to the investigation of tocotrienols' absorption.
7. Uncontrolled diabetes mellitus defined by an HbA1c of ≥ 7% in the last 3 months.
8. History of statin or other drug for cholesterol-control within 3 months before the start of the study.
9. Alcohol intake greater than "moderate" (one drink per day) or use of nonsteroidal anti-inflammatory drugs on a regular basis.
10. Cognitive impairment, depression or other medical/eating disorders, likely to move during the trial, lack of transportation, distance from the study site, or unavailable at sample collection times.
11. Smoking > 10 cigarettes/day.
12. Unwilling to accept randomization.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2022-10 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Serum bone resorption marker | baseline and after 12 weeks
  serum C-terminal cross-linked telopeptide of type I collagen, CTX Change from baseline CTX at 12 weeks. Investigators will also assess change from baseline CTX at 6 weeks.

SECONDARY OUTCOMES:
Serum bone formation marker | baseline, after 6 weeks, after 12 weeks
  serum N-terminal propeptide of type I collagen, PINP

OTHER OUTCOMES:
Oxidative stress marker | baseline, after 6 weeks, after 12 weeks
  8-hydroxy-2'-deoxyguanosine (8-OHdG) and urinary F2-isoprostanes (also called 8-iso-PGF2α)
Liver function test | baseline, after 6 weeks, after 12 weeks
  serum aspartate aminotransferase (ALT) and alanine aminotransferase (AST)
Quality of life Survey | baseline, after 6 weeks, after 12 weeks
  SF-36 survey (v2)
Serum tocotrienols concentrations | baseline, after 6 weeks, after 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Tech University Health Sciences Center, Lubbock, Texas, United States

REFERENCES:
- [Derived] Shen CL, Wang S, Yang S, Tomison MD, Abbasi M, Hao L, Scott S, Khan MS, Romero AW, Felton CK, Mo H. A 12-week evaluation of annatto tocotrienol supplementation for postmenopausal women: safety, quality of life, body composition, physical activity, and nutrient intake. BMC Complement Altern Med. 2018 Jun 28;18(1):198. doi: 10.1186/s12906-018-2263-0. PMID 29954374
- [Derived] Shen CL, Yang S, Tomison MD, Romero AW, Felton CK, Mo H. Tocotrienol supplementation suppressed bone resorption and oxidative stress in postmenopausal osteopenic women: a 12-week randomized double-blinded placebo-controlled trial. Osteoporos Int. 2018 Apr;29(4):881-891. doi: 10.1007/s00198-017-4356-x. Epub 2018 Jan 12. PMID 29330573
- [Derived] Shen CL, Mo H, Yang S, Wang S, Felton CK, Tomison MD, Soelaiman IN. Safety and efficacy of tocotrienol supplementation for bone health in postmenopausal women: protocol for a dose-response double-blinded placebo-controlled randomised trial. BMJ Open. 2016 Dec 23;6(12):e012572. doi: 10.1136/bmjopen-2016-012572. PMID 28011809